CLINICAL TRIAL: NCT02526199
Title: Protracted Mixture of Local Anesthetics for Major Foot and Ankle Surgery. A Randomized Double-blind, Controlled Study Comparing Bupivacaine-Epinephrine 0.5% Versus Bupivacaine-Epinephrine 0.5% With Dexamethasone
Brief Title: Protracted Mixture of Local Anesthetics for Major Foot and Ankle Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rasmus Wulff Hauritz (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor-Investigator, Rasmus Wulff Hauritz, Consultant Anesthesia, Kolding Sygehus
Organization: Kolding Sygehus (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2014-005383-14
Record Dates: First submitted 2015-08-11; First posted 2015-08-18 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Postoperative Pain
Keywords: Local anesthetics; Perineural nerve blocks; Perineurial Dexamethasone
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Epinephrine; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group BA (Active Comparator): Bupivacaine + Adrenaline Sciatic nerve block with Bupivacaine 0.5% + Epinephrine 5 microg/ml
  Interventions: Drug: Bupivacaine; Drug: Epinephrine
- Group BAD (Experimental): Bupivacine + Adrenaline + Dexamethasone Sciatic nerve block with Bupivacaine 0.5% + Epinephrine 5 microg/ml PLUS Dexamethsone 8 mg
  Interventions: Drug: Bupivacaine; Drug: Epinephrine; Drug: Dexamethasone

INTERVENTIONS:
Drug: Bupivacaine — Sciatic nerve block
  Other Names: Marcaine
Drug: Epinephrine — Adjuvant to perinerual block
  Other Names: Adrenaline
Drug: Dexamethasone — Adjuvant to perinerual block
  Other Names: Deaxagalene
  Arms: Group BAD

SUMMARY:
To extend the duration of peripheral nerve blockade after major foot and ankle surgery the investigators randomize the postoperative treatment with either perineurial sciatic nerve blocks with 0.5% Bupivacaine-Epinephrine with or without Dexamethasone.

ELIGIBILITY:
Inclusion Criteria:

* age > 17
* scheduled major foot and ankle surgery
* written informed consent
* fertile women in anti conceptive treatment
* fertile women not in anti conceptive treatment, but with negative urin-HCG on day of surgery

Exclusion Criteria:

* patients not able to understand or cooperate
* allergies to medicines involved
* daily buse of steroids
* daily use of opioids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-08; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Painfree period (time until first pain sensation in operated foot) | 48 hours
  Patients are closely monitored in the PACU until first pain sensation in the operated foot.

SECONDARY OUTCOMES:
Pain in the operated foot, measured on a numeric rating scale (0-10) | Every 30 minuttes from the patient enters the PACU to the nerve block wears of
  Pain score at rest, with the operated foot elevated on a pillow, ranging from 0 [no pain] to 10 [worst possible pain]
Sensibility score, measured with a hided tactile pinprick-sensation under the 3.rd toe on the operated foot | Every 30 minutes from the patient enters the PACU to the sensations core reach 2
  Sensitivy score measured on a 3 point scale 0 (no sensation) (impared sensation) 2 (full or normal sensation) compared to non-operated side
Total consumption of opioids during the length of stay | 48 hours
  A cummulative calculation of equipotente doses of oral milligrams of morphin during the length of stay
quality of sleep first night measured on a 3 point scale | hours
  Quality of sleep measured on the morning after operation. 0 (good sleep, no interruptions) by pain from operated foot) 1 (sleep, but interruption without pain) 2 (sleep but interrupted by pain from operated foot)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesia, Aarhus University Hospital, Aarhus, Region Midt, Denmark